CLINICAL TRIAL: NCT07011758
Title: Dynamic Treatment Regimes for Personalized Opioid Use Disorder Care
Brief Title: Dynamic Treatment Regimes for Opioid Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jason Brian Gibbons, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025p001360; K01DA061975 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dosage Forms; Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study uses a Sequential Multiple Assignment Randomized Trial (SMART) design. Participants are initially randomized in a 2x2 factorial structure in Week 1 to receive one of four treatment combinations. In Weeks 2-4, additional weekly treatment components are assigned based on participant response and predefined decision rules. This structure allows for evaluation of dynamic treatment regimens tailored to individual needs and evolving treatment response.
Masking Description: This is an open-label trial; no participants, providers, or investigators are masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Initial Intervention A + B (Experimental): Participants randomized to receive the combination of Intervention A and Intervention B in Week 1. Additional weekly interventions in Weeks 2-4 will be assigned based on participant response and dynamic treatment algorithms derived in Aim 1.
  Interventions: Drug: Medication for opioid use disorder; Behavioral: psychotherapy
- Initial Intervention A + D (Experimental): Participants randomized to receive the combination of Intervention A and Intervention D in Week 1. Subsequent treatment assignments in Weeks 2-4 follow adaptive treatment decision rules.
  Interventions: Drug: Medication for opioid use disorder; Behavioral: psychotherapy
- Initial Intervention C + B (Experimental): Participants randomized to receive the combination of Intervention C and Intervention B in Week 1. Adaptive treatment components are added weekly based on observed outcomes and predictive models.
  Interventions: Behavioral: psychotherapy
- Initial Intervention C + D (Experimental): Participants randomized to receive the combination of Intervention C and Intervention D in Week 1. Participants receive additional interventions in Weeks 2-4 based on dynamic treatment regimes developed in the modeling phase.
  Interventions: Behavioral: psychotherapy

INTERVENTIONS:
Drug: Medication for opioid use disorder — A medication treatment component delivered in Week 1 as part of a 2×2 factorial SMART design. The exact content (e.g., treatment modality or intensity) will be finalized based on model results from Aim 1, which identifies optimal dynamic treatment regimes.
  Arms: Initial Intervention A + B; Initial Intervention A + D
Behavioral: psychotherapy — A behavioral treatment component delivered in Week 1 as part of a 2×2 factorial SMART design. The exact content (e.g., treatment modality or intensity) will be finalized based on model results from Aim 1, which identifies optimal dynamic treatment regimes.

SUMMARY:
This study aims to develop and evaluate dynamic treatment regimes (DTRs) to improve personalized care for individuals with opioid use disorder (OUD). Using machine learning methods and longitudinal data from a national behavioral health provider, the investigators will identify optimal treatment sequences that minimize the risk of overdose and improve recovery outcomes. A pilot hybrid factorial SMART trial will be conducted to assess the feasibility and acceptability of implementing these personalized treatment decision rules in real-world clinical settings.

DETAILED DESCRIPTION:
This project supports the development and testing of dynamic treatment regimes (DTRs) for individuals with opioid use disorder (OUD), leveraging clinical and behavioral data from Discovery Behavioral Health and linked administrative records. In the first phase, multiple machine learning approaches (e.g., Q-learning, causal forests) will be used to estimate and validate DTRs that recommend tailored sequences of care based on patient characteristics and treatment response. The DTRs will be evaluated based on their ability to reduce fatal and non-fatal opioid overdose risk and hospital-based service use.

In the second phase, the investigators will conduct a pilot hybrid factorial Sequential Multiple Assignment Randomized Trial (SMART) to test the feasibility and acceptability of implementing the highest-performing DTR in a clinical setting. This pilot study will assess recruitment and retention, adherence to assigned treatment paths, and the practicality of integrating the DTR into routine care. The findings will inform a future full-scale trial aimed at improving personalized care for OUD and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with opioid use disorder (OUD)
* Receiving care at a participating Discovery Behavioral Health site
* Able to provide informed consent

Exclusion Criteria:

* Significant cognitive impairment or psychiatric instability that would prevent participation
* Current incarceration or involuntary commitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2028-07-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
CAT-SUD severity scores | 4 weeks
  Weekly Computerized Adaptive Test for Substance Use Disorder severity T-score. Scores range 0-100 (≈5-point precision). Higher scores indicate a greater SUD symptom burden/risk, while lower scores indicate fewer symptoms/lower risk. Prior validation studies have used <50 = low, 50-70 = intermediate, >70 = high severity/risk thresholds. Computerized Adaptive Test for Substance Use Disorder provides a dimensional severity score (not a diagnosis). Change is assessed week-to-week.
Retention in treatment | 4 weeks
  Whether participants remained engaged in behavioral health treatment through the end of the 4-week study period.
Patient and clinician satisfaction | 4 weeks
  Participant- and provider-reported satisfaction with the trial experience and procedures, assessed via standardized surveys.
Clinical fidelity to intervention protoco | Weekly over 4-week study period
  Fidelity of intervention delivery assessed via clinician checklists or independent fidelity ratings, evaluating adherence to protocol for each assigned treatment component.
Data completeness and consistency | Throughout the 4-week trial
  Proportion of participants for whom ethical standards are fully maintained (e.g., informed consent obtained, no reported violations).
  Proportion of participants for whom ethical standards are fully maintained (e.g., informed consent obtained, no reported violations).
  Proportion of EHR and survey data points with missing or inconsistent entries. Thresholds for success include <5% missingness or inconsistency.
Timeliness of EHR data entry | Weekly throughout the 4-week trial
  Proportion of EHR entries recorded within 48 hours of patient interaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Discovery Behavioral Health, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the study, including survey responses, CAT-SUD scores, and treatment assignments, will be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 1 year after study completion.
Access Criteria: equests will be reviewed by the principal investigator. Data will be shared through a secure data use agreement upon IRB approval and execution of a data-sharing agreement.